CLINICAL TRIAL: NCT07350538
Title: Pilot Exploratory Investigation Into DynaMAP Validation, Gut Microbiome Profiling, and Personalized Prebiotic Interventions for Alcohol Addiction Recovery
Brief Title: The Critical Link Between Gut Microbiome Dysfunction, Cravings and Relapse: RECLAIM-GUT TRIAL
Acronym: RECLAIM-GUT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Director, Principal Investigator, Clinical Professor, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LSC 25/ 431; AKT (Other Grant/Funding Number: UKRI); 10169630 (Other Grant/Funding Number: UKRI)
Record Dates: First submitted 2025-11-26; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Prospective interventional prebiotic pilot dietary clinical study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Following baseline analysis, each participant will receive a personalized prebiotic dietary formulation 1 or 2 or 3 as reported below (a nutritional supplement tailored to their microbiome profile as) to take daily for 60 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized prebiotic dietary Formulation 1 (Active Comparator): A nutritional prebiotic supplement tailored to their microbiome profile as to take daily for 60 days
  Interventions: Dietary Supplement: Personalized prebiotic dietary Formulation 1
- Personalized prebiotic dietary Formulation 2 (Active Comparator): A nutritional prebiotic supplement tailored to their microbiome profile as to take daily for 60 days
  Interventions: Dietary Supplement: Personalized prebiotic dietary Formulation 2
- Personalized prebiotic dietary Formulation 3 (Active Comparator): A nutritional prebiotic supplement tailored to their microbiome profile as to take daily for 60 days
  Interventions: Dietary Supplement: Personalized prebiotic dietary Formulation 3

INTERVENTIONS:
Dietary Supplement: Personalized prebiotic dietary Formulation 2 — Vitamin K Vitamin B1 Tryptophan Vitamin B6 Vitamin B5 Vitamin B9 Vitamin B3 Alpha-arabinooligosaccharides Ribose
  Arms: Personalized prebiotic dietary Formulation 2
Dietary Supplement: Personalized prebiotic dietary Formulation 3 — Lipoate Vitamin B9 Beta-glucosides Vitamin B5 Vitamin B7 Vitamin B6 Vitamin K Galactooligosaccharides Oligogalacturonate, Rhamnogalacturonides Fructooligosaccharides
  Arms: Personalized prebiotic dietary Formulation 3
Dietary Supplement: Personalized prebiotic dietary Formulation 1 — Chitobiose, Beta-glucosides Xylooligosaccharide Alpha-arabinooligosaccharides Fructooligosaccharides Ribose Oligogalacturonate, Rhamnogalacturonides
  Arms: Personalized prebiotic dietary Formulation 1

SUMMARY:
The human gut contains a vast community of microorganisms-including bacteria, viruses, and fungi-collectively known as the gut microbiota. This ecosystem co-evolves with humans and is shaped by diet, environment, and lifestyle. A balanced microbiota is essential for health, supporting immune function, regulating metabolism, and controlling intestinal inflammation. When this balance, or homeostasis, is disrupted, dysbiosis can occur, which has been linked to conditions such as inflammatory bowel disease, obesity, type 2 diabetes, cardiovascular disease, cancers, and neurological disorders. Evidence also shows that substance abuse can induce dysbiosis by altering microbial diversity, disrupting microbial composition, and reducing levels of key metabolites like short-chain fatty acids. Growing research on the gut-brain axis suggests that these microbial imbalances may influence mental health by affecting neurochemical signalling, contributing to disorders such as depression and anxiety. While synthetic drugs remain central to modern medicine and provide targeted, effective treatments, they often fall short when illnesses stem from disturbances within the microbial ecosystem. Because many conditions related to gut dysbiosis are not caused by a single malfunctioning molecule, traditional drugs may manage symptoms without restoring microbial balance. Some treatments, particularly broad-spectrum antibiotics, may even exacerbate dysbiosis by eliminating beneficial microbes. This has led to increasing interest in probiotics, prebiotics, and postbiotics. Probiotics are beneficial live microbes, prebiotics are non-digestible compounds that help these microbes grow, and postbiotics are their health-promoting byproducts. Although promising, these interventions are still considered supplements rather than formal medicines. Studying stool samples allows researchers to assess gut health by measuring bacterial and metabolic contents. Advances in this field require precise, efficient tools. Perseus Biomics' DynaMAP™ technology enables strain-level microbiome profiling. This study aims to validate DynaMAP™ against shotgun metagenomic sequencing and assess personalized prebiotic interventions based on individual microbiome profiles.

DETAILED DESCRIPTION:
A 60-day prospective, single-arm interventional pilot trial study in healthy adults who use alcohol moderately (6pints per week). A total of 20 participants will be invited to take part in this study. Open-label design (no blinding) since all participants will receive an active intervention (a personalized prebiotic) and there is no placebo/control group. The design features two main components within the same cohort: (1) a cross-sectional methodological comparison at baseline (comparing two lab methods on the same samples), and (2) a longitudinal intervention assessment (pre- vs post- supplementation within subjects).

ELIGIBILITY:
Inclusion criteria:

* Adults aged approximately 18-65 years
* Male or female
* Generally in good health, with no significant chronic illnesses
* Resident in the UK (to enable centralized ethics oversight and logistics)
* Able to re and understand English (for e-consent and study instructions)
* Mild to moderate alcohol consumption (more than 14 units or 6 pints per week)
* Willing to provide stool samples at the required time points
* Willing to take a daily prebiotic supplement for 60 days
* Has access to the internet and email for remote communication
* Able and willing to provide informed electronic consent

Exclusion criteria:

* Any known significant gastrointestinal disease (e.g., inflammatory bowel disease, celiac disease)
* Any major medical condition that could affect the gut microbiome or pose a health risk (e.g., immunocompromised conditions)
* Recent use of antibiotics (within the past 2-3 months)
* Recent regular use of probiotics or prebiotics (within approximately the past 4 weeks)
* Pregnant or breastfeeding women (pregnancy will be screened at enrolment, as the intervention is not tested during pregnancy and pregnancy itself alters the gut microbiome)
* Known allergies or intolerances to components likely used in the prebiotic formulation (e.g., certain amino acids)
* Use of special diets or medications that significantly alter gut microbiota (e.g., chronic laxative use, immunosuppressive therapy)
* Participation in another interventional clinical trial within the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome Taxonomic Composition | Baseline (Day 0) and Day 60 (end of prebiotic supplementation period)
  Change from baseline to Day 60 in gut microbiome taxonomic composition, measured as relative abundance of bacterial taxa from stool samples expressed as %
Microbial Functional Capacity - Fiber Fermentation | Baseline (Day 0) and Day 60 (end of prebiotic supplementation period)
  Change from baseline to Day 60 in predicted fiber fermentation capacity of the gut microbiome.Functional capacity score (arbitrary units derived from DynaMAP™ analysis)
Microbial Functional Capacity - Short-Chain Fatty Acid (SCFA) Production Potential | Baseline (Day 0) and Day 60 (end of prebiotic supplementation period)
  Change from baseline to Day 60 in predicted SCFA production potential of the gut microbiome in mmol/L

SECONDARY OUTCOMES:
Neurocognitive Performance - Attention | Baseline (Day 0) and Day 60 (end of prebiotic supplementation period)
  Change from baseline to Day 60 in attention performance, assessed using standardized computerized cognitive tasks administered via Inquisit.Task-based performance metrics (e.g., reaction time in milliseconds)
Neurocognitive Performance - Inhibitory Control | Baseline (Day 0) and Day 60 (end of prebiotic supplementation period)
  Change from baseline to Day 60 in inhibitory control performance. Task-based performance metrics
Self-Reported Mood and Psychological State | Baseline (Day 0) and Day 60 (end of prebiotic supplementation period)
  Change from baseline to Day 60 in self-reported mood and psychological state, assessed via validated questionnaires administered through Qualtrics.

CONTACTS AND LOCATIONS:
Overall Officials: ADELE COSTABILE, Study Director — University of Roehampton
Locations (1):
- University of Roehampton, School of Life and Health Sciences, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No